CLINICAL TRIAL: NCT06499389
Title: Randomized Controlled Trial Evaluating the Impact of Intensive, Instrumental and Early Respiratory Physiotherapy on Peak Expiratory Flow in Mechanically Ventilated Patients With ICU-acquired Muscle Weakness
Brief Title: Instrumental Respiratory Physiotherapy in Difficult-to-wean ICU Patients
Acronym: PHYSIO WEAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL23_1275; ID RCB (Other: 2024-A01433-44)
Record Dates: First submitted 2024-07-03; First posted 2024-07-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ventilator Weaning
Keywords: critical care; mechanical ventilation; ventilatory weaning; peak cough expiratory flow; cough strength; mechanical cough; extubation; reintubation; chest physiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive instrumental and early respiratory physiotherapy (Experimental): Patients in this arm will receive instrumental and intensive respiratory physiotherapy strategy from inclusion to day 7, 3 times a day, before and after extubation. Instrumental physiotherapy will be protocolized and cough strength and efficacy of bronchial secretions clearance will be evaluated
  Interventions: Procedure: Systematic and early intensive instrumental respiratory physiotherapy for patients undergoing difficult ventilatory weaning
- Protocolized standard-of-care respiratory physiotherapy (Active Comparator): Patients in this group will receive standardized and protocolized respiratory physiotherapy, i.e. 1 to 2 sessions of manual respiratory physiotherapy (not assisted by an instrumental technique) per day until the day of successful extubation, or until day 7 if necessary.
  Interventions: Procedure: Protocolized standard-of-care respiratory physiotherapy

INTERVENTIONS:
Procedure: Systematic and early intensive instrumental respiratory physiotherapy for patients undergoing difficult ventilatory weaning — Patients randomized to this group will receive 3 sessions per day of intensive early respiratory physiotherapy with instrumental techniques from randomization to day 7, before and after any extubation. The strategy will be applied until day 7 of randomization, regardless of the patient's status (intubated or not).
  Arms: Intensive instrumental and early respiratory physiotherapy
Procedure: Protocolized standard-of-care respiratory physiotherapy — Patients in this group will receive standardized and protocolized respiratory physiotherapy to reproduce the usual practices of non-expert centers,1 to 2 sessions of manual respiratory physiotherapy (not assisted by an instrumental technique) per day until the day of successful extubation, or until day 7 if necessary
  Arms: Protocolized standard-of-care respiratory physiotherapy

SUMMARY:
Difficult ventilatory weaning is associated with a 20% mortality rate. 40% of these patients will develop intensive care unit (ICU)-acquired neuromyopathy, associated with reduced cough strength and a 4-fold increase in the risk of reintubation. The objective measure of cough strength is peak expiratory flow (PEF). Instrument-assisted coughing is a respiratory physiotherapy technique capable of significantly increasing PEF in chronic neuromuscular patients and draining bronchial secretions.

The objective of the study is to determine whether an early, systematic, instrumental, intensive respiratory physiotherapy strategy in patients with difficult ventilatory weaning and ICU-acquired neuromyopathy significantly improves PEF immediately prior to extubation, compared with a conventional, protocolized management strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years or more, affiliated to a social security system
* Patients on invasive mechanical ventilation for 48 hours or more
* Failure of at least one mechanical ventilation weaning test (spontaneous breathing trial, SBT)
* First successful SBT on the day of eligibility assessment
* Medical Research Council (MRC) score < 48 and/or cough strength ≤ 2 on the 6-point Likert scale

Exclusion Criteria:

* Recent brain injury (< 3 months, stroke, cardiopulmonary arrest)
* Delirium tremens (Cushman score > 7)
* Chronic neuromuscular pathology
* Patient under continuous intravenous sedation
* Patient unresponsive to simple commands and Richmond Agitation and Sedation Scale (RASS) score < -2 or > +1
* FiO2: Inspired Oxygen Fraction> 50%, percutaneous, O2: oxygen saturation < 88%, positive end-expiratory pressure > 5 centimeter of water (cmH2O) or respiratory rate ≥ 35 min-1
* Vasopressor catecholamine at a dose > 0.5 μg/kg/min
* Tracheostomized patient
* Undrained pneumothorax
* Pulmonary emphysema (identified as antecedent in medical record)
* Uncontrolled hemoptysis
* Surgery < 3 months of esophagus and/or the ear, nose and throat (ENT) sphere
* Pregnancy or lactating
* Patient deprived of liberty by judicial or administrative decision
* Patient under guardianship or curatorship
* Patient already included in the same study or in another study sharing the same primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Unassisted peak expiratory cough flow (PECF) under mechanical ventilation during a voluntary coughing effort | At Hour 24
  PECF measured on the ventilator using its built-in flowmeter (PECF on unassisted coughing under mechanical ventilation). PECF is expressed in L/min.

SECONDARY OUTCOMES:
Unassisted PECF after disconnection from mechanical ventilation during a voluntary coughing effort | At Hour 24, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
  PECF measured by a spirometer without ventilation, either in intubated patients after disconnection from the ventilator, and in extubated patients by application of a naso-buccal mask connected to the spirometer. PECF is expressed in L/min.
Assisted PECF under mechanical ventilation | At Hour 24, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
  PECF measured by the spirometer during the application of mechanical (instrumental) cough assistance by connecting the spirometer between the intubation tube and the Cough Assist E70 in the intubated patient, or between the nasobuccal mask and the Cough Assist E70 in the extubated patient. PECF is expressed in L/min.
Semi-quantitative measurement of cough strength | At Hour 24, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
  Measurements of cough strength using a 6-level Likert scale (0-5) for intubated patients.
Semi-quantitative measurement of cough strength | At Hour 24, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
  Measurements of cough strength using a 4-level Likert scale (0-3) for extubated patients.
Semi-quantitative measurement of bronchial secretion quantity | At Hour 24, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7
  Measurements of bronchial secretion quantity using a 5-level Likert scale (0 to 4). The intensity of bronchial secretion quantity is graded semi-quantitatively by observing the quantity of secretions mobilized and/or present in the patient's airways.
Rate of hemodynamic instability episodes | At Hour 24 and after every respiratory physiotherapy session
  Number of physiotherapy sessions with mean arterial pressure < 65 mmHg. Hemodynamic instability is defined as the appearance of mottles, a mean arterial pressure < 65 mm Hg and requiring urgent intervention.
Ratio of arterial oxygen partial pressure to fractional inspired oxygen (O2) | At Hour 24, Day 7
  Ratios of arterial partial pressure in O2 to inspired fraction in O2 measured on the ventilator (P/F ratio). In extubated, non-ventilated patients, fraction of inspired oxygen (FiO2) will be estimated using the following formula: 〖fraction inspired oxygen (FiO)〗_2 (%)=21+O2 flow (in L/min)× 3. Partial oxygen pressure (PaO2) is measured on arterial blood gas.
Barotrauma complication rates | At Hour 24, Day 7
  Rate of barotraumatic complications. Thoracic (X-ray or computed tomography (CT) scan for pneumomediastinum and pneumothorax) or clinical examination (subcutaneous emphysema).
Reintubation rate | At Hour 24, Day 7
  Rate of reintubation
Number of days with invasive mechanical ventilation | Up to 60 days
  Time, in days, between inclusion and successful liberation from the ventilator
Ventilator-free days (VFD) | Up to 60 days
  Time alive and free from invasive mechanical ventilation. A VFD of 0 is adjudicated to patients who died over that period, even if they were liberated from mechanical ventilation.
Length of stay in intensive care unit | Up to 60 days
  Elapsed time, in days, between inclusion and ICU discharge

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service d'Anesthésie et Réanimation, Hôpital de la Croix Rousse, GHN, Lyon, France
  - Médecine Intensive - Réanimation, Hôpital de la Croix Rousse, Lyon
  - Département d'Anesthésie Réanimation - Médecine Intensive, Centre Hospitalier Lyon Sud, Lyon